CLINICAL TRIAL: NCT04637789
Title: Effectiveness of The Whole Body Vibration for Treating Sarcopenia in Hospitalized Patients Aged 80 Years and Older
Brief Title: The Whole Body Vibration for Sarcopenic Hospitalized Patients Aged 80+ Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuxiang Liang (Other)
Responsible Party: Sponsor-Investigator, Yuxiang Liang, Physiotherapist, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020（106）
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlled group (Other)
  Interventions: Behavioral: resistance training
- experimental group (Experimental)
  Interventions: Behavioral: the whole body vibration; Behavioral: resistance training

INTERVENTIONS:
Behavioral: the whole body vibration — most people stand on the platform with knees bent at about a 30-degree angle, while the surface beneath their feet vibrates an astounding 30 times per second.
  Arms: experimental group
Behavioral: resistance training — Resistance training is a form of exercise that improves muscular strength and endurance. During a resistance training workout, you move your limbs against resistance provided by your body weight, gravity,bands, weighted bars or dumbbells.

SUMMARY:
Resistance training have been recommended for sarcopenic patients. However, the whole body vibration training would further benefit for sarcopenic patients on the basis of resistance training remains unclear. The purpose of this study is to explore the effect of the whole body vibration training on improving the mobility of elderly patients with sarcopenia. The whole body vibration involves different frequencies that can improve muscle strength and keep aged upright, including the legs and core. These kinds of exercises can improve stability and help prevent falls.

ELIGIBILITY:
Inclusion Criteria:

* Sarcopenia defined by the Asia Working Group of Sarcopenia (AWGS)
* Agree to participant this study and sign the informed consent
* Aged 80 years or over

Exclusion Criteria:

* Patients who could not follow the training plan due to cognitive impairment, emotional problems or any other reasons;
* Severe heart and lung diseases;
* Renal insufficiency;
* Any type of tumor;
* Bedridden patients

Ages: 80 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
The change of activities of daily living | 3 Months
  Basic activities of daily living (BADL) assessed by Barthel Index

SECONDARY OUTCOMES:
The change of usual gait speed | 3 Months
The change of handgrip strength | 3 Months
The change of the score of Short Physical Performance Battery | 3 Months
The change of the score of Timed Up and Go test | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: ming Yang, Study Director — West China Hospital; jiaojiao Jiang, Study Director — West China Hospital
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China